CLINICAL TRIAL: NCT01008306
Title: Outcome After Pediatric Renal Transplantation: Cardiorespiratory Fitness, Cardiovascular Risk Factors and Quality of Life
Brief Title: Cardiovascular Risk Factors After Renal Transplantation in Children and Adults
Acronym: HENT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Red Cross (Other)
Responsible Party: Oslo University Hospital, Rikshospitalet HF, Rikshospitalet HF, department of pediatrics
Other Study IDs: S-07245b
Record Dates: First submitted 2009-11-03; First posted 2009-11-05 (Estimated); Last update posted 2009-11-05 (Estimated); Status verified 2009-11

CONDITIONS: Exercise Capacity; Physical Activity; Hypertension; Overweight and Obesity; Metabolic Syndrome
Keywords: Cardiorespiratory fitness; physical activity; hypertension; overweight and obesity; metabolic syndrome; Body composition
MeSH Terms: conditions — Motor Activity; Hypertension; Overweight; Obesity; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Freezing of serum and plasma from study participants
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Renal transplanted children and young adults: Renal transplanted children and adolescents (2-18yrs) transplanted between 1993-2006.
  Renal transplanted young adults aged 20-35 yrs old, transplanted from 1983 onwards.

SUMMARY:
Renal transplantation of children started in Norway in 1970.Since the beginning, >80% of renal transplants are provided from Living Donors(mainly parents), short pre-transplant dialysis time( median 4 months) and 50% of transplantations are performed before dialysis is needed.This gives good premises for graft survival and avoidance of detrimental effects of dialysis. However, renal transplanted children are subjected to an increased cardiovascular morbidity and mortality in adulthood due to consequences of chronic renal failure and immunosuppressive treatment.Cardiovascular death comprises 30-40% of death causes. In this cross-sectional study we evaluate cardiovascular risk factors in childhood- and also in young adults renal transplanted in childhood.

Focus is cardiorespiratory fitness using treadmill testing,24h BP measurements, anthropometrics including waist circumference,echocardiography,intima media thickness of carotids, glucose intolerance test.Participants are also requested to fill out physical activity recalls and Quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Transplanted after 1983, functioning graft

Exclusion Criteria:

* Patients in dialysis
* In part of the study concerning treadmill testing: Age<8 years, orthopedic limitations

Ages: 2 Years to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Renal transplanted children, adolescents and young adults transplanted in the period 1983-2006 in the same center (Oslo University Hospital, Rikshospitalet)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2007-06; Primary Completion 2010-06 (Estimated)

SECONDARY OUTCOMES:
other cardiovascular risk factors | 2007-2010
hypertension | 2007-2010
impaired glucose intolerance | 2007-2010
left ventricular hypertrophy, | 2007-2010

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital Rikshospitalet HF, Division of Pediatrics, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Sachs-Strommen K, Thorsteinsdottir H, Sakhi AK, Thomsen C, Lie A, Bjerre A, Lyche JL. Urinary levels and estimated daily intake of phthalates and phenols in kidney transplanted Norwegian children. Sci Total Environ. 2025 Oct 10;998:180251. doi: 10.1016/j.scitotenv.2025.180251. Epub 2025 Aug 21. PMID 40845701
- [Derived] Sitek JC, Tangeraas T, Bjerre A, Helsing P. The prevalence of skin disorders in Norwegian paediatric renal transplant recipients. Acta Derm Venereol. 2014 Jul;94(4):421-4. doi: 10.2340/00015555-1741. PMID 24287733